CLINICAL TRIAL: NCT00696202
Title: A Multicentre, Open Label, Uncontrolled Study of the Tolerance, Acceptability and Contraceptive Efficacy of Mirena 52 mg®, an Intra-uterine Levonorgestrel Device, During the First Year After Insertion Post-partum
Brief Title: Mirena Efficiency and Tolerability During the First Year of Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91295; 307702
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Medicated Intrauterine Devices; Contraception
Keywords: Mirena; Levonorgestrel; Intrauterine device; Efficacy; Tolerability; First year of use
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Mirena (BAY86-5028)

INTERVENTIONS:
Drug: Mirena (BAY86-5028) — Intrauterine levonorgestrel containing device (market product)

SUMMARY:
In this trial the efficacy and safety of Mirena was investigated during the first year of use

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 to 39 years who sought effective contraception during the post-partum period (i.e. insertion of the device between 6 and 12 weeks after parturition).

Exclusion Criteria:

* Standard exclusion criteria for use of intrauterine hormone devices

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2003-09; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Adverse event related to the product causing a subject to withdraw, or be withdrawn, from the study at any time up to 12 months from the insertion of Mirena | within 12 months after randomization

SECONDARY OUTCOMES:
General safety assessment | within 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Amiens, France